CLINICAL TRIAL: NCT06324799
Title: The Effect of Position Change Frequency on Hyperbilirubinemia in Term Infants Receiving Phototherapy
Brief Title: The Effect of Position Change Frequency on Hyperbilirubinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. prof, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/51
Record Dates: First submitted 2024-03-14; First posted 2024-03-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Newborn; Vitality; Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; newborn; Phototherapy
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Position group every 2 hours (Experimental): Newborns in the study group will change position (supine, prone, lateral) every 2 hours.
  Interventions: Other: phototherapy treatment
- Control group (No Intervention): Newborns in the control group will change position (supine, prone, lateral) every 6 hours.

INTERVENTIONS:
Other: phototherapy treatment — The newborns in the study group will be subjected to position changes (supine, prone, lateral) every 2 hours
  Arms: Position group every 2 hours

SUMMARY:
In our study, the effect of the frequency of position changes on hyperbilirubinemia in babies hospitalized in the Neonatal Intensive Care Unit and receiving phototherapy treatment will be investigated.

This study was planned as a single-center randomized controlled clinical trial to examine the effect of the frequency of position changes on the time it takes for hyperbilirubinemia to subside in babies receiving phototherapy treatment in the Neonatal Intensive Care Unit of Mersin City Training and Research Hospital.

Babies included in the study will be randomly divided into two groups by randomization method. While the babies in the study group will be subjected to position changes (supine, prone, lateral) every 2 hours, the same procedure will be applied to the control group every 6 hours. All newborns included in the study were treated with the Unitest (Blue angel) LED Phototherapy device, which is used as standard in the neonatal intensive care unit, at a distance of 25-40 cm, at a wavelength of 425-475 nm, at 45 watts, at 50/60 Hz. Phototherapy will be applied unidirectionally. During phototherapy, only the perineal area of the babies will be covered with a reduced diaper, and their eyes will be covered with a three-layer, cotton, black eye patch that transmits 99.5% of ultraviolet rays. During phototherapy sessions, the total serum bilirubin level of the patient is checked; Phototherapy will be continued until it falls below the threshold value in the Bhutani nomogram, which is evaluated according to postnatal days and risk factors. The descriptive characteristics of the babies included in the study and their total bilirubin and hematocrit values before the start of phototherapy will be recorded on the form prepared by the researchers. After phototherapy begins, position changes will be made every two hours for babies in the experimental group and every six hours for babies in the control group until the total serum bilirubin value falls below the phototherapy threshold value in the Bhutani nomogram.

Bilirubin levels will be measured and recorded by venous measurement at the sixth hour and the 24th hour, and this process will be continued regularly until the bilirubin value decreases to the normal range. This practice is performed routinely in the clinic and will not be considered specific to the study.

DETAILED DESCRIPTION:
This study was planned as a single-center randomized controlled clinical trial to examine the effect of the frequency of position changes on the time it takes for hyperbilirubinemia to subside in babies receiving phototherapy treatment in the Neonatal Intensive Care Unit of Mersin City Training and Research Hospital.

Randomization and Masking: Randomization will be achieved by randomly and equally distributing patients who meet the sample selection criteria to 2 groups (group 1 study group and group 2 control group) through a computer program. Randomization will also be stratified according to the feeding style of the babies, as breast-fed babies may affect the duration of phototherapy. Stratified randomization will be performed according to whether the babies are fed with breast milk or formula.

(http://www1.assumption.edu/users/avadum/applets/RandAssign/GroupGen.html).

Babies included in the study will be randomly divided into two groups by randomization method. While the babies in the study group will be subjected to position changes (supine, prone, lateral) every 2 hours, the same procedure will be applied to the control group every 6 hours. All newborns included in the study were treated with the Unitest (Blue angel) LED Phototherapy device, which is used as standard in the neonatal intensive care unit, at a distance of 25-40 cm, at a wavelength of 425-475 nm, at 45 watts, at 50/60 Hz. Phototherapy will be applied unidirectionally. During phototherapy, only the perineal area of the babies will be covered with a reduced diaper, and their eyes will be covered with a three-layer, cotton, black eye patch that transmits 99.5% of ultraviolet rays. During phototherapy sessions, the total serum bilirubin level of the patient is checked; Phototherapy will be continued until it falls below the threshold value in the Bhutani nomogram, which is evaluated according to postnatal days and risk factors. The descriptive characteristics of the babies included in the study and their total bilirubin and hematocrit values before the start of phototherapy will be recorded on the form prepared by the researchers. After phototherapy begins, position changes will be made every two hours for babies in the experimental group and every six hours for babies in the control group until the total serum bilirubin value falls below the phototherapy threshold value in the Bhutani nomogram.

Bilirubin levels will be measured and recorded by venous measurement at the sixth hour and the 24th hour, and this process will be continued regularly until the bilirubin value decreases to the normal range. This practice is performed routinely in the clinic and will not be considered specific to the study.

In both groups, babies will start phototherapy in the prone position, and the patients will continue to be fed 8 times a day, at 3-hour intervals, as the routine of the neonatal intensive care unit. Babies will be fed by turning off phototherapy for a maximum of 15 minutes, thus minimizing phototherapy interruption. Care will be taken not to exceed this period for babies who are breastfed by their mothers.

Data Collection Tools

Baby Identification Information Form: The form includes descriptive characteristics of the babies included in the study; It includes questions about their gender, mode of birth, birth weight, gestational age, Apgar score, weight, bilirubin level and hematocrit level.

Bhutani Nomogram: Each bilirubin value must be interpreted according to the "bilirubin nomogram" prepared according to the baby's age in hours. The use of the nomogram according to postnatal age allows monitoring the course of repeated bilirubin values and predicting the baby who will later develop hyperbilirubinemia. This scale, known as the "Bhutani nomogram" and has been widely used since 1999, will be used in our study.

Evaluation of Data The analysis of the data obtained from the research will be carried out in the SPSS 22.0 statistical package program. The statistical significance level was determined as 0.05. Kolmogrow-Smirnov will be used in the normality analysis of dependent variables. Chi-square and comparison of means tests will be used to determine the similarity of the groups. In comparing between and within groups averages, appropriate parametric or non-parametric tests will be used, depending on whether the distribution is normal. In addition, at the end of the research, whether the study has been conducted with a sufficient sample size will be tested with post-hoc power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Born after 37 weeks of gestation, receiving treatment at Mersin City Training and Research Hospital Neonatal Intensive Care Service,
* There is an indication for phototherapy treatment in the phototherapy nomogram, where the total serum bilirubin value is evaluated according to the patient's postnatal day and risk factors,
* Postnatal 1-15. on the day,
* Patients whose families approve the informed consent form.

Exclusion Criteria:

* Older than the 15th postnatal day,
* There is an indication for exchange transfusion in the blood exchange curve, where the total serum bilirubin value is evaluated according to the patient's day and risk factors,
* Having a major anomaly or disease detected antenatally,
* Patients with comorbid diseases such as perinatal asphyxia, bronchopulmonary dysplasia, intraventricular hemorrhage, necrotizing enterocolitis, congenital heart disease and similar diseases will not be included in the study.

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Bhutani Nomogram | 1 day
  Each bilirubin value must be interpreted according to the "bilirubin nomogram" prepared according to the baby's age in hours. The use of the nomogram according to postnatal age allows monitoring the course of repeated bilirubin values and predicting the baby who will later develop hyperbilirubinemia. This scale, known as the "Bhutani nomogram" and has been widely used since 1999, will be used in our study.

SECONDARY OUTCOMES:
bilirubin level | 1 day
  bilirubin level in blood
hematocrit levels | 1 day
  hematocrit value in blood

CONTACTS AND LOCATIONS:
Overall Officials: Çağla Tarcan, Principal Investigator — Mersin University
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] American Academy of Pediatrics, Clinical Practice Guideline, Subcommittee on Hyperbilirubinemia. Management
- [Result] Karen Marcdante & Robert M. Kliegman & Abigail M. Schuh. 2023 Nelson Essentials of Pediatrics 9th edition. 2022. p. 953-60.
- [Result] Ovalı F., Dağoğlu T. Neonatoloji. İndirekt Hiperbilirubinemi. 3. Baskı İstanbul: Nobel Tıp Kitabevleri Tic. Ltd. Şti.; 2018. p. 959-84.
- [Result] Bhethanabhotla S, Thukral A, Sankar MJ, Agarwal R, Paul VK, Deorari AK. Effect of position of infant during phototherapy in management of hyperbilirubinemia in late preterm and term neonates: a randomized controlled trial. J Perinatol. 2013 Oct;33(10):795-9. doi: 10.1038/jp.2013.54. Epub 2013 Jun 6. PMID 23743672
- [Result] Thukral A, Deorari A, Chawla D. Periodic change of body position under phototherapy in term and preterm neonates with hyperbilirubinaemia. Cochrane Database Syst Rev. 2022 Mar 2;3(3):CD011997. doi: 10.1002/14651858.CD011997.pub2. PMID 35235686
- [Result] Shinwell ES, Sciaky Y, Karplus M. Effect of position changing on bilirubin levels during phototherapy. J Perinatol. 2002 Apr-May;22(3):226-9. doi: 10.1038/sj.jp.7210678. PMID 11948386
- [Result] Akkuzu, A. (2021). Hiperbilirubinemi tanısı ile yenidoğan yoğun bakım ünitesinde yatan bebeklerin beslenme şekilleri ile hastanede kalış süreleri arasındaki ilişki (Master's thesis, İstanbul Medipol Üniversitesi Sağlık Bilimleri Enstitüsü).
- [Result] Donneborg ML, Knudsen KB, Ebbesen F. Effect of infants' position on serum bilirubin level during conventional phototherapy. Acta Paediatr. 2010 Aug;99(8):1131-4. doi: 10.1111/j.1651-2227.2010.01885.x. Epub 2010 Jun 2. PMID 20528799
- [Result] Lee Wan Fei S, Abdullah KL. Effect of turning vs. supine position under phototherapy on neonates with hyperbilirubinemia: a systematic review. J Clin Nurs. 2015 Mar;24(5-6):672-82. doi: 10.1111/jocn.12712. Epub 2014 Oct 16. PMID 25319831
- [Result] Chen CM, Liu SH, Lai CC, Hwang CC, Hsu HH. Changing position does not improve the efficacy of conventional phototherapy. Acta Paediatr Taiwan. 2002 Sep-Oct;43(5):255-8. PMID 12607480